CLINICAL TRIAL: NCT04496258
Title: Investigating the Neural Systems That Support the Beneficial Effects of Positive Emotion on Stress Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kateri McRae, Associate Professor, University of Denver
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1606445; 2R15MH106928-02A1 (NIH)
Record Dates: First submitted 2020-07-16; First posted 2020-08-03 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Behavior
Keywords: cognition; reappraisal
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive VR Scene (Experimental): Participants will explore a virtual reality (VR) environment of a beach scene. Participants will be randomly assigned (between subjects) to beach or office scene. VR will be presented on an Occulus Rift device.
  Interventions: Behavioral: Positive Emotion Induction
- Neutral VR Scene (Experimental): Participants will explore a virtual reality (VR) environment of a neutral office scene. Participants will be randomly assigned (between subjects) to beach or office scene. VR will be presented on an Occulus Rift device.
  Interventions: Behavioral: Neutral Emotion Induction

INTERVENTIONS:
Behavioral: Positive Emotion Induction — Participants are expected to have a positive emotional response to the more positive beach scene.
  Arms: Positive VR Scene
Behavioral: Neutral Emotion Induction — Participants are expected to have a neutral emotional response to the neutral office scene.
  Arms: Neutral VR Scene

SUMMARY:
For this study, community participants visited the PI's psychophysiology lab for a single experimental session. In this study, participants completed a brief mood measure, followed by a task training in which a research assistant described and gave examples of cognitive reappraisal in response to negative images. Participants were then randomly assigned to positive or neutral emotion induction conditions, delivered by virtual reality. Then, participants completed an event-related, picture-based cognitive reappraisal task for 23 minutes. Following the task, participants once again responded to a mood measure, completed post-task questionnaires (individual difference measures) and answered a series of questions regarding the task they completed, including difficulty of regulation, or any images that were personally relevant.

The investigators predicted that the positive emotion induction would result in powerful effects on self-reported emotion, which may or may not interact with the cognitive reappraisal condition.

DETAILED DESCRIPTION:
For the studies, participants were recruited via paper and electronic flyers on campus and in the surrounding communities. Interested participants were screened via phone, email and/or web form to assess eligibility according to criteria listed elsewhere. If participants qualified, they were be invited to complete a single laboratory session in the PI's lab.

Once arriving at the laboratory, participants completed the consent process, in which a research assistant trained in ethical principles regarding human subjects research answered any questions about the consent form and verbally reinforced the key rights of the participants outlined there. Once both parties were satisfied, the consent form was signed.

Participants sat with a trained research assistant/experimenter who gave an overview of the entire session, and then began training for the cognitive reappraisal task. The training took 10-15 minutes. During the training, the experimenter offered several possible reappraisals of negative images and allowed the participants to offer their own as well, providing encouragement and feedback. During this training, the experimenter also went over the method of responding (using the VR equipment). Participants were reminded during training that they may stop the experiment at any point if the pictures are too upsetting.

Immediately following task training, participants will made a general mood rating using the mDES. Then, they were randomly assigned to a positive or neutral mood induction, to be delivered via the VR headset for three minutes. Participants were encouraged to explore the VR environment, which was either a positive (beach scene) or neutral (office scene). The VR environment was implemented using a headset with integrated audio. After the VR exploration, participants made a rating of their current positive and negative affect in the VR environment. Then, participants completed the reappraisal task in the VR environment. The task took approximately 23 minutes.

Finally, participants completed post-task individual difference measures.

ELIGIBILITY:
Inclusion Criteria:

* Community members ages 18-55
* Fluent in English
* Without present psychotic symptoms

Exclusion Criteria:

* None

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kateri McRae, Ph.D., Principal Investigator — University of Denver
Locations (1):
- The University of Denver, Frontier Hall, Denver, Colorado, United States

REFERENCES:
- [Derived] Kako N, Waugh CE, McRae K. The Future of Immersive Mood Induction in Affective Science: Using Virtual Reality to Test Effects of Mood Context on Task Performance. Affect Sci. 2023 Sep 12;4(3):570-579. doi: 10.1007/s42761-023-00213-1. eCollection 2023 Sep. PMID 37744975

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive VR Scene | Neutral VR Scene
Started | 49 | 50
Completed | 47 | 49
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive VR Scene | Neutral VR Scene | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 49 | 96
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.98 (4.33) | 19.08 (1.45) | 19.5 (3.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 17 | 15 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 40 | 45 | 85
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 30 | 37 | 67
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 47 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: Mood Ratings (Pos)
Description: Before putting on the VR headset and at the end of the experiment, participants used the modified Differential Emotions Scale (mDES; Fredrickson, 2013; Izard, 1977) to rate their current mood. We defined the mDES as a mood measure because it was intended to measure participants' current mood absent of a stimulus intended to evoke an emotional response (Rosenberg,1998). The mDES consists of 20 questions and is comprised of two sub-scales for positive and negative emotions with 10 questions for each subscale respectively. Scales are comprised of averaging all positive scores together and all negative scores together. In our study, participants were asked to rate their current experience of all 20 emotions on a five-point Likert Scale (1 - not at all to 5 - Extremely). Minimum socre = 1, maximum score = 5. Higher scores indicate higher levels of positive/negative mood.
Time Frame: Baseline, and post-reappraisal task
Population: Several pre-registered exclusion criteria were applied prior to data analysis including: lack of understanding of the task (N = 5), missing more than 25% of trial level data (N = 8). Additional participants were excluded due to a corrupted data file (N =1) and mixing up the positive and negative ratings (N = 1), and outlier scores greater than 3 standard deviations above/below the mean for most outcome measures (N= 1). This left usable data for a total of 80 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
units on a scale
  Baseline Positive | 1.34 (.57) | 1.04 (.53)
  Post-Task Positive | .96 (.6) | .83 (.54)
  Baseline Negative | .81 (.34) | .77 (.51)
  Post-Task Negative | .71 (.42) | .72 (.49)

2. Primary Outcome: Means of Self-reported Emotion Ratings
Description: The mean of each negative and positive emotion score were calculated post-reappraisal task. Higher scores indicate higher positive and negative emotions. The scale for both positive and negative was 1 - 9 where 1 was not positive at all/not negative at all and 9 was very positive/very negative. The minimum score was 1 and the maximum score was 9.
Time Frame: During the reappraisal task, individual ratings for each picture were taken immediately after viewing the image. The mean rating across all images was computed after the experiment was complete.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
units on a scale
  Negative emotion rating in response to viewing neutral images | 2.68 (.84) | 2.75 (1.13)
  Positive emotion rating in response to viewing neutral images | 5.09 (1.81) | 4.35 (1.81)
  Negative emotion rating in response to viewing negative images | 5.33 (1.49) | 5.90 (1.12)
  Positive emotion rating in response to viewing negative images | 3.5 (1.63) | 2.81 (1.14)
  Negative emotion rating in response to reappraising negative images | 4.14 (1.46) | 4.24 (1.38)
  Positive emotion rating in response to reappraising negative images | 4.44 (1.58) | 3.86 (1.37)

3. Primary Outcome: Mood Induction Ratings
Description: After the VR induced mood induction, and prior to starting the reappraisal task participants rated their positive and negative emotions on a 1-9 scale, where 1 is not at all and 9 is extremely.
Time Frame: Pre-reappraisalTask
Population: In addition to the exclusion criteria discuss above, certain participants appeared to miss the time window they had to make their rating selection.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 40 | 36
units on a scale
  Positive Rating | 7.38 (1.56) | 4.81 (2)
  Negative Rating: number analyzed (Participants) | 33 | 25
  Negative Rating | 1.45 (.83) | 2.52 (1.61)

4. Secondary Outcome: Debriefing of Instructions
Description: Following the VR task, participants were asked to report the task instructions in their own words. The first questions asked participants to reiterate the instructions they were given for the cognitive reappraisal task (for example: "What were you instructed to do during the 'LOOK' trials?") This is a fill in the blank question and there are no right or wrong answers. All participants' responses are viewed to ensure understanding of the task instruction. There are no scores to report for this measure. Rather this, outcome serves more as a comprehension check than an actual analysis of interest.
Time Frame: Post-reappraisal task
Population: Participants who completed and had full data for the in-person experiment.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 47 | 49
Participants | 41 | 39

5. Secondary Outcome: Task Difficulty
Description: The next batch of questions asked the participants questions about the difficulty of the task. The questions asked were: "How difficult was it to follow the 'LOOK' instruction?" And: "How difficult was it to follow the 'DECREASE' instruction?" Participants will be rating the level of difficulty on a scale of 1 to 7 with 1 being "not difficult at all" to 7 being "very difficult". There are no right or wrong answers to this question. The range of scores is 1-7.
Time Frame: Post-reappraisal task
Population: Participants who completed and had full data for the in-person experiment and passed all other exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
units on a scale
  Look Difficulty Rating | 2.41 (1.55) | 2.4 (1.53)
  Decrease Difficulty Rating | 4.55 (1.9) | 4.5 (1.9)

6. Secondary Outcome: Number of Participants With Full Task Compliance
Description: Participants were asked about self-reported task compliance. For example, one question asked "What percentage of the time were you able to follow the "LOOK" instruction?" The participants were rating their self-compliance for each task from 0% (non-compliant) to 100% (fully compliant). There are no right or wrong answers to this question and these responses are more descriptive/exploratory. They are not used in any specific analyses. The number of participants analyzed below indicates the number of participants that were fully compliant across both conditions.
Time Frame: Immediately after the reappraisal task
Population: Participants who completed and had full data for the in-person experiment and passed all other exclusion criteria.
Measure: Number; unit: participants
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
participants | 41 | 39

7. Secondary Outcome: Number of Participants Reviewed for Possible Prior Experience With the Reappraisal Task and/or Task Images
Description: Participants were asked whether they have any experience with reappraisal or the specific images presented in the task. The first question asked "Have you ever been trained to change your emotions by changing the way you think (in therapy, or in another experiment, or anywhere else)?" Participants can choose "Yes" or "No" for this question. The participant will have to extrapolate if they have changed their emotions before using a fill in the blank. The next question asked"Have you ever seen any of these exact emotional images before?" If participants answered yes, they were once again asked to extrapolate which images they have seen and what emotional response was generated by these images using a fill in the blank option. These are descriptive and not used in any formal analyses. The number of participants analyzed below indicates the the number of participant responses we reviewed.
Time Frame: Post-reappraisal task
Population: Participants who completed and had full data for the in-person experiment and passed all other exclusion criteria.
Measure: Number; unit: participants
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
participants | 41 | 39

8. Secondary Outcome: DWECK-E (Theries of Emotion Scale)
Description: The theories of emotion scale was developed for use by Maya Tamir, Oliver P. John, Sanjay Srivastava, and James J. Gross in 2007, based on Carol Dweck's Implicit Theories of Intelligence scale (Dweck, 1999). It's used to measure beliefs about the malleable nature of emotion on a scale of 1 (strong disagree) to 5 (strongly agree) where higher scores indicate stronger agreement with the belief. There are 4 items, 2 of which are reverse coded. Scores are taken by averaging the response items. The minimum score is 1 and the maximum range is 5.
Time Frame: Post-reappraisal task
Population: Participants who completed and had full data for the in-person experiment and passed all other exclusion criteria.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale | 3.59 (.81) | 3.46 (.70)

9. Secondary Outcome: The Big Five Inventory-10 (BFI-1)
Description: A 10 item self-report scale that is designed to measure the big five personality traits (extraversion, agreeableness, conscientiousness, neuroticism, and openness) on a scale of 1-5 where higher values indicate higher indication of the personality trait. Certain individual items are reversed scored on this measure. The subscales in our data were calculated using averages to produce a score. The possible range for each subscale reported included a minimum value of 1 and a maximum value of 5.
Time Frame: Post-reappraisal task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale
  Extraversion | 3.27 (1.14) | 2.99 (.94)
  Agreeableness | 3.84 (.96) | 3.42 (.96)
  Conscientiousness | 3.6 (.96) | 3.65 (.97)
  Neuroticism | 3.28 (1.06) | 3.27 (1.02)
  Openness | 3.63 (.78) | 3.64 (.97)

10. Secondary Outcome: Brief Resilience Scale
Description: The BRS is a self-report measure that assesses the ability to bounce back or recover from stress on a 1-5 scale. Higher scores indicate higher levels of resilience.
Time Frame: Post-reappraisal task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale | 2.83 (.69) | 2.69 (.62)

11. Secondary Outcome: Satisfaction With Life Scale
Description: A 5-item scale designed to measure global cognitive judgments of one's life satisfaction (not a measure of either positive or negative affect). Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. Higher scores indicate higher levels of satisfaction. The scale is summed to produce a score, and the possible range of scores is 5-35.
Time Frame: Post-reappraisal task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale | 22.32 (6.25) | 21.31 (5.74)

12. Secondary Outcome: The Igroup Presence Questionnaire (IPQ)
Description: The Igroup Presence Questionnaire (IPQ) is a self-report scale for measuring the sense of presence experienced in a virtual environment (VE). It contains three subscales that assess aspects of presence: spatial presence, involvement, and experience realism. Higher scores indicate higher sense of presence. Items were rated on a scale of 0 to 6 and items for each subscale are averaged to get each subscale core. The Range for all subscales are 0-6.
Time Frame: Post-reappraisal task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale
  Spatial Presence | 3.73 (.73) | 3.58 (1.15)
  Involvement | 3.79 (1.4) | 3.21 (1.25)
  Experience Realism | 2.39 (.89) | 2.43 (1.17)

13. Secondary Outcome: Brief Cope
Description: The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. Sub-scales are reported. Higher scores indicate higher use of the coping strategy. he Brief COPE is comprised of 14 scales, each of which assesses the degree to which a respondent utilizes a specific coping strategy. The scales are: Active Coping, Planning, Positive Reframing, Acceptance, Humor, Religion, Using Emotional Support, Using Instrumental Support, Self-Distraction, Denial, Venting, Substance Use, Behavioral Disengagement, Self-Blame. Items are rated on a 4-point Likert scale, ranging from 1 - "I haven't been doing this at all" to 4 - "I've been doing this a lot." Each of the scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum).
  Total scores for each sub scales are calculated by summing the items. There is no overall total score.
Time Frame: Post-reappraisal task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale
  Self-Distraction | 4.66 (1.24) | 4.49 (1.32)
  Active Coping | 5.39 (1.53) | 5.59 (1.57)
  Denial | 2.59 (1) | 3.08 (1.71)
  Substance Use | 3.37 (1.93) | 3.41 (1.80)
  Emotional Support | 5.37 (1.73) | 5 (2)
  Instrumental Support | 5.2 (1.86) | 4.74 (1.76)
  Behavioral Disengagement | 3.07 (1.57) | 3.03 (1.09)
  Venting | 4.05 (1.22) | 3.85 (1.44)
  Positive Reframing | 5.29 (1.33) | 4.92 (1.58)
  Planning | 5.29 (1.63) | 5.49 (1.64)
  Humor | 4.95 (1.64) | 5.08 (1.75)
  Acceptance | 5.63 (1.67) | 6.13 (1.34)
  Religion | 3.32 (1.97) | 3 (1.56)
  Self-Blame | 4.93 (1.59) | 5.15 (1.65)

14. Other Pre Specified Outcome: Depression Trait Differences
Description: The participants were given the Beck's Depression Inventory(BDI-II) which measures symptoms of depression and were used to examine any between-subjects trait differences. The BDI-II is a 21 self-report measure looking at symptoms of depression with ratings falling between 0 and 3 (0 being "not at all" and 3 would indicate experiencing these symptoms on a constant basis). There are no subscales. Higher scores indicate higher levels of depressive symptoms. Scores range from 0 - 63
Time Frame: Post-reappraisal task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale | 12.37 (9.32) | 13.73 (7.45)

15. Other Pre Specified Outcome: Emotional Regulation Trait Differences
Description: The Emotion Regulation Questionnaire (ERQ) looks at methods of regulating emotions and will be used to examine any between-subjects trait differences. The ERQ is a 10-item self-report questionnaire assessing the use of two strategies to alter emotions: cognitive reappraisal and expressive suppression. The scale is rated on a 7-point Likert scale with 1 being "strongly disagree" and 7 being "strongly agree". Six items are categorized as using cognitive reappraisal while four of the items assess expressive suppression. Higher scores indicate higher use of the emotion regulation strategies. The scale scores were computed by taking the average of the items included in each sub scale. The possible range for each sub scale is 1-7
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive VR Scene | Neutral VR Scene
Number analyzed (Participants) | 41 | 39
score on a scale
  Cognitive Reappraisal Scale | 4.99 (.96) | 4.81 (.89)
  Expressive Suppression Scale | 3.35 (1.33) | 4.01 (1.27)

ADVERSE EVENTS:
Time Frame: The duration of the in-person experiment (approximately 90 minutes)
Description: Potential risks included mild psychological discomfort from the stress tasks and negative emotional pictures, but not above levels normally experienced in daily life. To mitigate the risks of psychological discomfort, we use only procedures that have been established in previous studies to pose no more than the minimal psychological discomfort participants. RAs were trained to check in with participants regularly and reminded participants they could stop the study at any time.
Arm/Group | Positive VR Scene | Neutral VR Scene
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT04496258/Prot_SAP_000.pdf